CLINICAL TRIAL: NCT04863651
Title: Do Patient's Adult Attachment Style Correlate With Pain Post Cesarean Delivery?
Brief Title: Attachment Predicts Post Cesarean Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: WREM114262
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Cesarean Section Complications; Attachment Disorder; Post Operative Recovery
Keywords: Cesarean; Cesarean Section; Attachment Style; Revised Adult Attachment Style; Post Cesarean Pain; Post Cesarean Recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Securely Attached Parturients: Parturients who have a secure attachment style according to the Revised Adult Attachment Scale (Collins, 1996)
- Insecurely Attached Parturients: Parturients who have an insecure attachment style according to the Revised Adult Attachment Scale (Collins, 1996)

SUMMARY:
The Adult Attachment Style (AAS) is a questionnaire designed to measure how an adult generally feels in their close personal relationships. The questionnaire has two main axes of measurements - avoidance and anxiety, that gives rise to four different categories of attachment styles. Women's attachment styles have been shown to be correlated to pain during labour, but not after. No study has analyzed whether attachment styles are correlated to the pain after cesarean section. This study will assess correlation between the AAS score, and pain after elective cesarean section. Additionally, this study aims to clarify the correlation between attachment scale and overall quality of recovery after cesarean section as defined by a recently validated tool, the ObsQoR10.

DETAILED DESCRIPTION:
Overall recovery after cesarean section is difficult to measure and must consider several factors that may influence recovery. The ObsQoR10 is a recently validated tool that provides an overall picture of post cesarean recovery using pain, functional milestones, and emotional needs1. One of the factors that may influence recovery post operatively is a person's Adult Attachment Style (AAS).

AAS refers to how a person "generally feels in close relationships in their lives" and is prevalent in literature in the context of chronic pain. AAS has been shown to be correlated to patients' psychological stress2, self reported pain intensity and even the prevalence of chronic pain conditions like fibromyalgia3. In a cohort of patients with chronic pain, securely attached individuals were less likely to report disability due to pain, depressive symptoms and perceived negative spouse responses in comparison to securely attached individuals4. Another cohort showed that patients were characterized as fearful avoidant were more likely to catastrophize their pain and exhibit activity avoiding behaviours5.

Literature on AAS in the context of pain experienced by parturients is not as well characterized. Costas-Martins et al showed that insecurely attached women experience more pain during labour6. Costas-Martins et al include in their cohort a number of cesarean patients but do not consider them separately. To date there has not been a study investigating whether the AAS of parturients undergoing cesarean section is correlated to their perceived pain.2

While pain is an important clinical outcome, overall recovery as measured by the ObsQoR10 may present a more complete clinical picture of the predictive power of a person's AAS. Our study aims to characterize whether parturients' AAS is correlated with their overall recovery post cesarean section as well as pain.

ELIGIBILITY:
Inclusion Criteria:

i. English Speaking ii. Elective Cesarean Sections iii. ASA 3 or lower iv. Singleton Pregnancy v. Between 37-40 weeks gestation

Exclusion Criteria:

i. Patient Refusal ii. History of chronic pain condition, currently on medication iii. Diagnosed General Anxiety Disorder iv. Diagnosed substance use disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 65 English speaking parturients undergoing elective cesarean section at Victoria Hospital's Obstetrical Care Unit will be approached prior to their scheduled operation.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 24 hours
  Pain score from 0-10, measured at 24 hours post-operative

SECONDARY OUTCOMES:
ObsQoR10 Score | 24 hours
  Total score on the ObsQoR10 tool, a quality of recovery tool post cesarean section. Collected at 24 hours post-operative.
Total Opioid Consumption first 24h | 24 hours
  Total consumption of opioids by the patient in the first 24 hours post-operative, including the time at which additional opioid analgesia was first requested by the patient.
First Occurrence of Nausea | 24 hours
  The first time the patient reports feeling nauseous within the first 24 hours post-operative.
First Occurrence of Vomiting | 24 hours
  The first time the patient reports feeling vomiting within the first 24 hours post-operative.
First Occurrence of Pruritis | 24 hours
  The first time the patient reports feeling vomiting within the first 24 hours post-operative.
First Occurence of Sedation | 24 hours
  The first time the patient reports feeling sedated within the first 24 hours post-operative.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Sebbag, MD, Principal Investigator — Western University
Locations (1):
- Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Study data will only be linked to a research number which will be correlated with identifying information on a master list paper copy only accessible to the members of this study.
  Data will not be shared with researchers whom are not included in this study.

REFERENCES:
- [Background] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408
- [Background] Lee SS, Rim HD, Won SH, Woo J. Avoidant Insecure Attachment as a Predictive Factor for Psychological Distress in Patients with Early Breast Cancer: A Preliminary 1-Year Follow-Up Study. Psychiatry Investig. 2018 Aug;15(8):805-810. doi: 10.30773/pi.2018.06.07. Epub 2018 Aug 9. PMID 30086610
- [Background] Penacoba C, Perez-Calvo S, Blanco S, Sanroman L. Attachment styles, pain intensity and emotional variables in women with fibromyalgia. Scand J Caring Sci. 2018 Jun;32(2):535-544. doi: 10.1111/scs.12477. Epub 2017 Sep 8. PMID 28885733
- [Background] Andrews NE, Meredith PJ, Strong J, Donohue GF. Adult attachment and approaches to activity engagement in chronic pain. Pain Res Manag. 2014 Nov-Dec;19(6):317-27. doi: 10.1155/2014/838954. Epub 2014 Oct 22. PMID 25337857
- [Background] Costa Martins JM, da Silva CF, Pereira M, Martins H, Oliveira C, Puga A, Coelho R, Tavares J. Women's attachment as a predictor of pain during labour and post-delivery: a prospective observational study. Acta Med Port. 2014 Nov-Dec;27(6):692-9. doi: 10.20344/amp.4960. Epub 2014 Dec 30. PMID 25641282
- [Background] Suso-Ribera C, Sullivan MJL, Suso-Vergara S. Pain Intensity Is Not Always Associated with Poorer Health Status: Exploring the Moderating Role of Spouse Personality. Pain Res Manag. 2018 Sep 26;2018:7927656. doi: 10.1155/2018/7927656. eCollection 2018. PMID 30356426